CLINICAL TRIAL: NCT07357623
Title: Surufatinib Plus Standard Chemotherapy Versus Surufatinib Monotherapy in Patients With Pulmonary Neuroendocrine Tumors: a Randomized, Controlled, Open-label Study
Brief Title: Surufatinib Combined With Chemo Versus Surufatinib in the Treatment of Pulmonary Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Chief physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-NEN113
Record Dates: First submitted 2025-08-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Neuroendocrine Tumor
Keywords: surufatinib, NET, Typical carcinoid, Atypical carcinoid
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib Combined With Standard chemotherapy (Experimental): Standard chemotherapy included either Capecitabine combined with Temozolomide or Etoposide plus Carboplatin
  Interventions: Drug: Surufatinib Combined With Standard chemotherapy
- Surufatinib (Active Comparator)
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib Combined With Standard chemotherapy — Surufatinib: 250mg , qd, po, Q4W Capecitabine: 75mg/m2, bid, po, D1-D14, Q4w Temozolomide: 150mg-200mg/m2, qd, po, D10-D14, Q4W or Surufatinib: 250mg , qd, po, Q3W Etoposide: 100mg/m2, IV, D1-D3, Q3W Carboplatin: AUC=5, IV, D1, Q3W
  Arms: Surufatinib Combined With Standard chemotherapy
Drug: Surufatinib — Surufatinib: 300mg, qd, po
  Arms: Surufatinib

SUMMARY:
The goal of this clinical trial is to investigate if chemotherapy works with surufatinib to treat pulmonary neuroendocrine tumors. It will also learn about the safety of this combination regimen. The main questions it aims to answer are:

Does chemotherapy combined with surufatinib could bring more survival benefits (ie. higher response rate or longer survival time) for patients with pulmonary neuroendocrine tumors? Is this combination regimen safe?

Researchers will compare chemotherapy plus surufatinib with surufatinib monotherapy to see if this combination regimen works to treat pulmonary neuroendocrine tumors.

Participants will:

Take chemotherapy(Etoposide+Carboplatin, EC or Capecitabine+Temozolomide, CAPTEM) plus surufatinib or surufatinib monotherapy every 3 or 4 weeks as a cycle.

Visit the clinic once every cycle for checkups and tests. Tumor assessment is performed every 2 cycles. Treatment will continued until disease progression, death, intolerable toxicity, or withdrawn.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of this study and voluntarily sign the informed consent form;
2. 18-75 years old (including cut-off value), male or female;
3. Patients must have at least one measurable lesion (RECIST 1.1);
4. Histologically or cytologically confirmed pulmonary neuroendocrine tumor (typical or atypical carcinoid) [at least one neuroendocrine immunohistochemistry marker (CD56, CgA, Syn) definitively positive on the basis of morphological features of neuroendocrine tumors];
5. Patients who have not received systemic therapy in the past (Note: neoadjuvant or adjuvant chemotherapy is allowed in the early stage, and if disease progression/recurrence occurs ≥ 6 months after the end of neoadjuvant/adjuvant last therapy, it can also be included);
6. ECOG PS 0-1 (PS 0-2 for amputees);
7. Expected survival ≥ 12 weeks;
8. Blood test (without blood transfusion within 14 days) 1) Absolute neutrophil value ≥1.5×109/L, platelet ≥ 100×109/L, hemoglobin ≥9g/dL; 2) Liver function tests (AST and ALT≤2.5×ULN, total bilirubin≤1.5×ULN; AST and ALT ≤5×ULN) if liver metastases are present; 3) Renal function (serum creatinine ≤1.5×ULN, creatinine clearance (CCr) ≥60ml/min);
9. Male or female patients of childbearing potential voluntarily use effective contraceptive methods, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. during the study and within 6 months of the last study medication. All female patients will be considered of childbearing potential unless the female patient is naturally postmenopausal, has undergone artificial menopause, or has undergone sterilization (e.g., hysterectomy, bilateral adnextomy, or radioactive ovarian irradiation, etc.).

Exclusion Criteria:

1. Patients who have received surufatinib or other anti-angiogenic drugs in the past;
2. Received approved or investigational systemic anti-tumor therapy within 4 weeks before enrollment, including: chemotherapy, any form of radiotherapy, biological immunotherapy, targeted therapy, etc.;
3. Participated in other domestic drug clinical trials that have not been approved or marketed within 4 weeks before enrollment and received corresponding trial drug treatment;
4. Undergoing any surgery or invasive treatment or operation within 4 weeks before enrollment that affects wound healing (except for intravenous catheterization, puncture and drainage, etc.);
5. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) >1.5× ULN;
6. Clinically significant electrolyte abnormalities judged by the investigator;
7. Presence of hypertension that cannot be controlled by medication, as prescribed as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
8. Patient currently has any disease or condition that affects drug absorption, or patient cannot take surufatinib orally;
9. Patients currently have active gastric and duodenal ulcers, ulcerative colitis and other gastrointestinal diseases or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation as determined by the investigator;
10. Patients with obvious evidence or history of bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months, hematemesis, black feces, blood in the stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attack) within 12 months;
11. Significant clinically significant cardiovascular disease, including but not limited to the following: acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure New York Heart Association (NYHA) grade >2; ventricular arrhythmias requiring medication; LVEF (left ventricular ejection fraction) < 50%;
12. Other malignant tumors within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
13. Active or uncontrolled serious infection:

1) Known human immunodeficiency virus (HIV) infection; 2) Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., HBV DNA positive (>1×104 copies/mL or >2000 IU/ml); 3) Known hepatitis C virus infection (HCV) with positive HCV RNA (>1×103 copies/mL), or other hepatitis, cirrhosis; 14. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects who have been previously treated for brain metastases may be enrolled provided that the patient's disease is clinically stable for at least 2 weeks and there is no evidence of new or enlarging brain metastases and steroids are off 3 days prior to administration of study drug. According to this definition, stable brain metastases should be determined prior to the first dose of study drug. Subjects with asymptomatic brain metastases (i.e., no neurological symptoms, no need for corticosteroids, and no lesions >1.5 cm) may be enrolled, but require regular imaging of the brain as a site of disease; 15. Patients with persistent toxicity caused by any previous anti-tumor therapy that has not recovered to grade ≤2, but have any grade of alopecia and lymphopenia are allowed to participate in this study; 16. Pregnant (positive pregnancy test before medication) or breastfeeding; 17. Received blood transfusion therapy, blood products and hematopoietic factors such as albumin and granulocyte colony-stimulating factor (G-CSF) within 14 days before enrollment; 18. The investigator believes that the subject has any clinical or laboratory abnormalities or other reasons that are not suitable for participation in this clinical study; 19. Those who showed urine protein ≥ 2 and had a quantitative of > 1.0g in 24 hours;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR)(RECIST1.1) | From date of enrollment to the end of treatment, an average of 1.5 years
  The incidence of confirmed complete response or partial response

SECONDARY OUTCOMES:
Disease control rate (DCR)(RECIST1.1) | From date of enrollment to the end of treatment, an average of 1.5 years
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Progression-free Survival (PFS) (RECIST1.1) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  A duration from the date of randomization to disease progression or death of any cause.
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Duration from the date of randomization to the date of death due to any cause
4-month PFS rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 months
  Proportion of patients who did not develop disease progression (or death from any cause) at 4 months from the date of randomization

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai chest hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No